CLINICAL TRIAL: NCT04114500
Title: The Association Between Serum Estradiol and Progesterone on the Same Day of FET and the Pregnancy Outcome
Brief Title: The Association Between Serum E2 and P on the Day of FET and the Pregnancy Outcome
Acronym: FET
Status: Completed | Type: Observational
Sponsor: Al Baraka Fertility Hospital (Other)
Responsible Party: Principal Investigator, Dr. Kamal Rageh, doctor , medical director, Al Baraka Fertility Hospital
Other Study IDs: KAMAL
Record Dates: First submitted 2019-09-22; First posted 2019-10-03 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Frozen Embryo Transfer
Keywords: Estradiol; FET; IVF; Progesterone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum estradiol and progesterone — blood sample for measuring serum estradiol and progesterone level on the same day of FET

SUMMARY:
The outcomes of frozen embryo transfer (FET) have substantially improved over the last decade, due to the improvements in the cryopreservation process, Artificial endometrial preparation is typically accomplished by the administration of estradiol (E2) supplementation and exogenous progesterone (P) in order to transform the endometrium into a secretory one, mimicking a natural cycle , The current study aims to determine the association, if any, between serum E2 and P levels, measured same day of FET, and pregnancy outcome

DETAILED DESCRIPTION:
Study design a retrospective cohort study for 402 FET cycles which will be conducted in Al- Baraka Fertility Hospital, Manama, Bahrain, between April 2018 and May 2019. The trial registration number for the study is (NCT04114500), and it was approved by our ethical committee Study population

* Inclusion criteria were women who underwent FET, were age below 40 yrs., body mass index (BMI) below 30 kg/m2, patients who underwent FET treatment using the endometrial preparation was initiated with oral estradiol valerate, the endometrial thickness was no less than 8 mm on the day when P was administrated; with normal endometrial ultrasound imaging and euploid pre-genetically tested embryos;
* Exclusion criteria were chromosomal and genetic disorders, age> 40 years, BMI > 35 , abnormal ultrasonogram of uterine cavity (acquired or congenital) and abnormal embryos not suitable for transfer.

Study protocol Endometrial preparation in frozen embryo transfer (FET) briefly, patients received treatment with 2 mg/8h E2 (Estrofem, Novo Nordisk) for 12-14 days, Endometrial thickness was evaluated with transvaginal sonography. When endometrial thickness reached 8 mm or greater and was trilaminar in appearance, patients were initiated on both vaginal micronized P (Crinone gel, Merck) and oral P (Duphastone, Abott) treatment at 200 mg/8h. P4 was given as supplementation because normal ovarian steroid production and the ovarian follicular-to-luteal transition were suppressed with estradiol. A depot GnRH agonist was administered in the midluteal phase of the preceding cycle at clinician's discretion. On the early morning of day 5 of P treatment, the same day of FET, a blood sample was obtained and immediately analyzed. Hormone determinations of E2 and P were performed. Then, embryo transfer of the pre-genetically tested euploid embryos was performed under ultrasound guidance. 12 days later pregnancy test was assessed, 4 weeks after FET date ultrasound will be scheduled to check the viability and clinical pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent frozen-thawed embryos transfer treatment
* the endometrial preparation was initiated with oral estradiol valerate
* the endometrial thickness was no less than 8 mm on the day when P was administrated;
* normal endometrial ultrasound imaging
* euploid pre-genetically tested embryos

Exclusion Criteria:

* age> 40 years
* BMI > 35
* abnormal ultrasonogram of uterine cavity
* abnormal embryos not suitable for transfer

Ages: 22 Years to 40 Years | Sex: Female
Age Groups: Adult
Study Population: Patients undergoing IVF/FET were recruited from April 2018 to September 2019.
Sampling Method: Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-05 (Actual)

PRIMARY OUTCOMES:
Pregnancy rate | 2 weeks
  B-hCG
clinical pregnancy rate | 4 weeks
  positive fetal heart beat

CONTACTS AND LOCATIONS:
Locations (1):
- Al-BARAKA FERTILITY HOSPITAL, Manama, Adliya, Bahrain

IPD SHARING:
Plan to Share IPD: Undecided